CLINICAL TRIAL: NCT05710770
Title: Double-blinded, Randomized, Sham-controlled Trial of Immunoadsorption (IA) in Patients With Chronic Fatigue Syndrome (CFS) Including Patients With Post-acute COVID-19 CFS (PACS-CFS)
Brief Title: Immunoadsorption in Patients With Chronic Fatigue Syndrome Including Patients With Post-COVID-19 CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Harald Pruess, Director of the Department of Experimental Neurology, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA-PACS-CFS; 01EP2201 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2023-01-31; First posted 2023-02-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-04

CONDITIONS: ME/CFS; Post-COVID ME/CFS
Keywords: Post-COVID Syndrome; Long COVID; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome | interventions — Plasmapheresis

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunoadsorption (Active Comparator): Immunoadsorption will be conducted with the TheraSorb LIFE 21 apheresis system in combination with the TheraSorb-Ig omni 5 adsorber over a period of 9-12 days: each participant will receive five immunoadsorption cycles treating 2.0 - 2.5 patient's plasma volumes every other day. Initial pilot studies have demonstrated this dose finding to be effective and well tolerated (Scheibenbogen et al., 2018; Tolle et al., 2020). The immunoapheresis material will be provided by the Miltenyi company at the beginning of the study.
  Concerning the high effectiveness of immunoadsorption therapy in patients with other neuroimmunological diseases and the invasiveness of a sham-apheresis, a 2:1 randomization was chosen in order to ensure that more patients will receive a verum IA treatment.
  Interventions: Device: Immunoadsorption
- Sham-apheresis (Sham Comparator): To have identical conditions to the immunoadsorption, sham apheresis will also be conducted with the TheraSorb LIFE 21 apheresis system over a period of 9-12 days: each participant will receive five sham cycles. For the sham apheresis, a TheraSorb LIFE 21 unit with blocked Ig adsorbers and without regeneration of the adsorbers during the treatment will be used, ensuring that the patient and the investigator are blinded. The study nurses applying the treatment (a specific person only in charge of the patient during the treatment) cannot be blinded.
  Interventions: Device: Immunoadsorption

INTERVENTIONS:
Device: Immunoadsorption — IA is a well-established, safe interventional therapy broadly applied for different indications. Medical complaints of the TheraSorb Ig apheresis system are rare and none led to a long-term impairment of the patient's health. In most treatments, the patients do not report any side effects. The Ig omni adsorbers specifically remove antibodies. Other components of the blood, except for an unspecific loss of plasma during the treatment, are not removed. Main adverse effects can occur due to the necessity of a Shaldon catheter and include accidental puncture of carotid artery. The procedure is performed under sonographic control and a chest-x-ray is performed afterwards to ensure integrity of lungs.

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of repeated immunoadsorption intervention in patients with chronic fatigue syndrome (CFS) including patients with post-acute COVID-19 CFS (PACS-CFS).

The main questions it aims to answer are: (1) Does repeated immunoadsorption relieve fatigue and/or other symptoms associated with CFS and PACS-CFS? (2) Is repeated immunoadsorption safe and tolerable in this patient population? What are the side effects of repeated immunoadsorption, and how common are they?

Participants will be asked to participate for approx. 32 weeks (8 months). After screening, participants will receive assigned intervention of either five immunoadsorption treatments (with Ig adsorber) every other day over 10 days or matching sham treatments (without Ig adsorber), followed by a 6-month follow-up period with three ambulatory visits. Every participant will undergo trial outcome, safety, and monitoring assessments.

The results of this study will provide information on whether repeated immunoadsorption can alleviate symptoms associated with CFS and PACS-CFS, as well as insights into the pathophysiological processes in this condition, which in turn can help to develop new and effective therapies.

DETAILED DESCRIPTION:
Myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) is a severely debilitating condition with a varying prevalence of 0.3 - 3% and markedly restricts activity and function of patients. They experience severe fatigue even after minimal exercise or mental activity, together with a myriad of further symptoms such as cognitive impairment, poor sleep quality, muscle and joint pain, or headache. With the pandemic situation, ME/CFS related to post-acute COVID-19 syndrome (PACS) is becoming a raising issue. According to the WHO (in February 2022), there are more than 423 million confirmed cases of COVID-19 worldwide and a large proportion of patients discharged from hospital are suffering from persistent symptoms (Carfi et al., 2020; Davis et al., 2020).

The etiology and the mechanisms leading to the typical chronic course of ME/CFS or the pathophysiology of PACS are not fully understood. There is increasing evidence that a post-viral autoimmune reaction with the presence of autoantibodies targeting different neuronal tissues is involved in the pathogenesis.

This is a double-blinded, randomized, sham-controlled immunoadsorption (IA) study in patients with chronic fatigue syndrome (CFS) including patients with CFS related to post-acute COVID-19 syndrome (PACS-CFS). Primary endpoint of the study is clinical improvement 3 months after the completion of immunoadsorption (IA) quantified using the change from baseline of the Chalder Fatigue Scale (range 0-33). Patients are randomized 2:1 in order to provide therapy to as many patients as possible. During the screening period, all patients are tested for the presence of autoantibodies in blood and cerebrospinal fluid (CFS). A comprehensive characterization by CFS specific questionnaires, quality of life questionnaires (PROMIS), cognitive and neuropsychological testing (MOCA, CANTAB) is performed, and each patient is offered to receive an optional cranial MRI before and after immunoadsorption. Depending on the clinical phenotype, electromyography and pulmonary function testing will be done. We use established hand strength and finger tapping devices as well as an accelerometer to objectify clinical improvement. Patients are hospitalized for 9-12 days receiving IA 5 times every other day. Directly after completion of IA as well as at month 1, 3 and 6 there are followup visits.

The study will help to better understand disease mechanisms and thereby allow (hopefully biomarker associated) characterization of patients benefitting from such a costly but safe and often highly efficient therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of all genders ≥18 <65 years at time of informed consent
* Diagnosed ME/CFS according to Canadian consensus criteria (CCC) 2003 including patients with PACS-CFS at screening with Bell Score ≥20 and ≤50
* Detection of at least one kind of autoantibodies measured during screening (among others antineuronal-, ß2-adrenergic-receptor-, muscarine-receptorantibodies) in serum or CSF

Exclusion Criteria:

* Comorbidity bearing risk that patient might not tolerate treatment as judged by investigator including among others:

  * malignant disease within the last 5 years
  * clinically meaningful laboratory abnormalities
  * moderate to severe renal insufficiency
  * cardiac insufficiency with an LVEF lower than 40%, uncontrolled cardiac arrhythmia, severe coronary heart disease
  * severe Hypercoagulability
* Acute or severe psychiatric disease
* Current indispensable medication with ACE inhibitors
* Fatigue duration for ≥5 years
* Presence of other conditions or differential diagnosis better explaining the symptoms of the patient than the suspected ME/CFS
* Ongoing immunosuppressive therapy
* Active/acute infectious diseases like TBC, HIV, CMV, EBV, HBV, HBC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Improvement in physical and mental fatigue as measured by the Chalder Fatigue Scale | 3 months after completion of immunoadsorption or sham apheresis
  The Chalder Fatigue Scale measures the extent and severity of tiredness and has been used in multiple randomized trials of behavioral interventions in patients with ME/CFS. Each of the 11 items is answered on a 4-point scale with an overall score ranging from 0 (asymptomatic) to 33 (maximum symptomology). Intra-patient change in physical and mental fatigue from baseline to month three will be documented as indexed by the Chalder Fatigue Scale.

SECONDARY OUTCOMES:
Sustained improvement quantified by the Chalder Fatigue Scale | 10 days, 1 month, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  Intra-patient change in physical and mental fatigue from baseline to follow-up points will be documented.
Verification of safety and tolerability of immunoadsorption in this patient population | 1 day, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  Number of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and discontinuation due to TEAEs
Improvement in severity of symptoms of chronic fatigue syndrome (CFS) as measured by the Fluge score | 1 month, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  The Fluge score uses a visual analogue scale ranging from 1 to 10 (1 = no symptom, 10 = very severe symptom) to assess 32 self-reported CFS symptoms including fatigue, pain, cognitive, and other CFS-related symptoms. Intra-patient change in Fluge score from baseline to follow-up points will be documented.
Improvement in physical function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | 1 month, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  The Short Form 36 Health Survey (SF-36) is an established and widely used health-related quality of life measure. The Physical Function (PF) domain asks patients to report limitations on ten mobility activities, such as walking specified distances, carrying groceries, and bathing or dressing. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, i.e., severe disability) to 100 (no health restrictions). An intra-patient change in SF-36-PF from baseline to follow-up points will be documented.
Improvement in functional disability as measured by the Bell disability scale | 1 month, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  The Bell disability scale is a standard assessment in ME/CFS that evaluates functional ability in adult ME/CFS patients. Eleven statements describe patient status such as level of symptoms at rest, level of symptoms with exercise, activity level, and ability to perform work, travel and self care. Its score ranges from 0 (bedridden) to 100 (no symptoms). Intra-patient change in Bell score from baseline to follow-up points will be documented.
Improvement in fatigue quantified by post exertional malaise (PEM) questionnaire | 1 month, 3 months, and 6 months after completion of immunoadsorption or sham apheresis
  The PEM questionnaire determines frequency (from 0 to 20 points, higher scores equate to greater frequency), severity (from 0 to 20 points, higher scores equate to greater severity), and length (from 0 to 6 points, higher scores equate to longer duration) of PEM. Intra-patient change in PEM score from baseline to follow-up points will be documented.
Improvement in muscle fatigue measured by the repetitive hand grip strength test (HGS) | 10 days, 3 months, and optional 6 months after completion of immunoadsorption or sham apheresis
  Intra-patient change in hand grip strength (HGS) from baseline to follow-up points.
Improvement in symptoms of autonomic dysfunction as measured by the Composite Autonomic Symptom Score (COMPASS-31) | 10 days, 3 months, and optional 6 months after completion of immunoadsorption or sham apheresis
  The Composite Autonomic Symptom Score (COMPASS-31) is a refined, internally consistent, and markedly abbreviated quantitative measure of autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, applies a much-simplified scoring algorithm, and is suitable for widespread use in autonomic research and practice. It evaluates six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains. The score ranges from 0 (no symptoms) to 100 (strong autonomic dysfunction). Intra-patient change in autonomic dysfunction from baseline to follow-up points will be documented as indexed by the COMPASS-31.
Improvement in symptoms of autonomic dysfunction by measuring blood pressure and heart rate regulation with the Schellong Test | 10 days, 3 months, and optional 6 months after completion of immunoadsorption or sham apheresis
  The Schellong Test is a test for circulatory function. The patient is required to stand for 10 to 20 min, during which time the blood pressure is measured continuously. A fall of systolic pressure of 20 mm Hg or more indicates poor circulatory function. Intra-patient change in Schellong Test from baseline to follow-up points will be documented.
Improvement in neurocognitive functions as measured by the Montreal Cognitive Assessment (MoCA) | 3 months and 6 months (only if requested by the investigator) after completion of immunoadsorption or sham apheresis
  MoCA is a sensitive and validated cognitive screening tool to test subjects quickly and accurately for mild cognitive impairment, irrespective of etiology. A person can gain a maximum of 30 points, and professionals consider a score of 26 or above to be normal. A score of 25 points or less may indicate some degree of cognitive impairment (18-25 = mild cognitive impairment, 10-17 = moderate cognitive impairment, fewer than 10 points = severe cognitive impairment). Intra-patient change in neurocognitive functions at month 3 and at month 6 (if required by the investigator) after IA completion compared to baseline.
Improvement in neurocognitive functions as measured by the symbol digit modalities test (SDMT) | 3 months and 6 months (only if requested by the investigator) after completion of immunoadsorption or sham apheresis
  The SDMT (oral version) detects cognitive impairment in less than five minutes and will be used to assess change in cognitive function over time. SDMT is a validated and established measure of cognition in multiple sclerosis capturing impairments such as processing speed and working memory, visual search and scanning and oculomotor functioning. Patients are provided a sheet with nine symbols, each paired with a number on top of the page. The remainder of the page consists of a randomized, sequential assortment of these symbols. Participants are asked to verbally respond with the number that corresponds with each symbol. The final score is the correct number of substitutions in 90 s (range 0 to 110, higher score = higher neurocognitive function). Intra-patient change in neurocognitive functions at month 3 and at month 6 (if required by the investigator) after IA completion compared to baseline.
Improvement in quality of life (QoL) as measured by the PROMIS questionnaire | 3 months and optional 6 months after completion of immunoadsorption or sham apheresis
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS measures can be used with the general population and with individuals living with chronic conditions. Intra-patient change in PROMIS score from baseline to follow-up points will be documented.
Changes in biomarkers of autoimmune activity | 3 months after completion of immunoadsorption or sham apheresis
  Intra-patient changes in biomarkers of autoimmune activity (autoantibody titers against neurotransmitter receptors; among others ß2-adeno-receptor- and muscarine- receptor-antibodies) in blood and optional in cerebrospinal fluid at month 3 after IA completion compared to baseline.
Changes in biomarkers of inflammation | 3 months and 6 months after completion of immunoadsorption or sham apheresis
  Intra-patient change in biomarkers of inflammation (CRP, ferritin, MBL, white blood cell count, complement factors, cytokines, immunoglobulin level and subtype) in blood at month 3 and 6 after IA completion compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Prüß, Prof., MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Scheibenbogen C, Loebel M, Freitag H, Krueger A, Bauer S, Antelmann M, Doehner W, Scherbakov N, Heidecke H, Reinke P, Volk HD, Grabowski P. Immunoadsorption to remove ss2 adrenergic receptor antibodies in Chronic Fatigue Syndrome CFS/ME. PLoS One. 2018 Mar 15;13(3):e0193672. doi: 10.1371/journal.pone.0193672. eCollection 2018. PMID 29543914
- [Background] Tolle M, Freitag H, Antelmann M, Hartwig J, Schuchardt M, van der Giet M, Eckardt KU, Grabowski P, Scheibenbogen C. Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Efficacy of Repeat Immunoadsorption. J Clin Med. 2020 Jul 30;9(8):2443. doi: 10.3390/jcm9082443. PMID 32751659
- [Derived] Pressler H, Machule ML, Ufer F, Bunger I, Li LY, Buchholz E, Werner C, Beraha E, Wagner F, Metz M, Burock S, Bruckert L, Franke C, Wilck N, Kruger A, Reshetnik A, Eckardt KU, Endres M, Pruss H. IA-PACS-CFS: a double-blinded, randomized, sham-controlled, exploratory trial of immunoadsorption in patients with chronic fatigue syndrome (CFS) including patients with post-acute COVID-19 CFS (PACS-CFS). Trials. 2024 Mar 7;25(1):172. doi: 10.1186/s13063-024-07982-5. PMID 38454468

DOCUMENTS (1):
  • Statistical Analysis Plan: SAP (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05710770/SAP_000.pdf